CLINICAL TRIAL: NCT01442779
Title: Clinical Trial of Low Dose Oral Interferon Alpha in Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: Ainos, Inc. (f/k/a Amarillo Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00190
Record Dates: First submitted 2009-09-23; First posted 2011-09-29 (Estimated); Results first posted 2011-09-29 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Interstitial; Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Interferon alpha
MeSH Terms: conditions — Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Interstitial; Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Interferon alpha oral lozenge — dose form - oral lozenge dose - 150 International Units (IU) frequency - 3 times a day duration - at least 1 year

SUMMARY:
The purpose of this study is to determine the possible efficacy of low dose, orally administered interferon alpha in subjects with Idiopathic Pulmonary Fibrosis (IPF).

DETAILED DESCRIPTION:
This is a pilot study to determine if oral administration of low doses of Interferon alpha might be effective in treating Idiopathic Pulmonary Fibrosis (IPF). This is a disease that damages the lungs leading to marked decreases in the quality of life and death within 3-5 years after diagnosis. The cause is unknown. The standard treatment has for some time been steroids such as prednisone or prednisolone because of their anti-inflammatory actions, but there is little evidence that steroids either improve the condition, prevent further deterioration or improve life expectancy. Additionally, they have many side effects.

In this disease, normal cells are damaged for unknown reasons and replaced by a type of scar. This scar tissue prevents the easy movement of oxygen from the lungs into the blood, making it difficult for the patient to perform normal activities. With progression, which usually occurs rapidly, patients require supplemental oxygen to perform even simple tasks.

Interferons are chemicals normally produced in the body and the rate of their production has been shown to be reduced in the lungs of patients with IPF. They are involved in regulating the activity of the immune system which may play a role in initiating the damage to the lungs in IPF and they also can inhibit the activity of the cells that form the scar tissue. Our hypothesis is that treating patients with interferon might prevent damage to additional normal tissue and prevent the formation of additional scar tissue. This would prevent progression, improve the quality of life and extend the expected life span if successful. Another study has been ongoing in which IPF patients have been given injections of large doses of another type of interferon. This treatment regimen is expensive and side effects have been fairly frequent.

In contrast, we are treating IPF patients with low doses of interferon administered orally. The interferon is taken three times per day by letting a lozenge dissolve in the mouth. These low doses have been shown to produce effects in patients with other diseases and they produce very few side effects. If side effects occur, they usually are not severe and go away quickly. Those reported most commonly by other subjects have been headaches, nausea, rashes, respiratory infections, sore throat or diarrhea. No one has had to stop taking the medicine because of the side effects. The medicine is provided free of charge.

This study has been going on for about 5 years. The subjects are given the same tests that they receive as part of their standard of care. These include chest x-rays, High Resolution CT scans, pulmonary function tests and some blood tests. They are done before starting interferon alpha, and, depending on the test, are repeated at 3-, 6-, 9- or 12 month intervals. In addition subjects are asked to complete questionnaires on the quality of life, cough history and a dyspnea index at each visit.

ELIGIBILITY:
Inclusion Criteria:

* The only subjects to be included in this study are those diagnosed with Idiopathic Pulmonary Fibrosis with diagnosis based on the criteria published by the American Thoracic Society in the International Consensus Statement.

  1. Exclusion of other known causes of interstitial lung disease.
  2. Abnormal pulmonary function studies.
  3. Bibasilar reticular abnormalities with minimal ground glass opacities on HRCT scan.
  4. Biopsy or lavage showing no features supporting alternative diagnosis.
  5. Patient older than 50 years of age.
  6. Insidious onset of otherwise unexplained dyspnea on exertion.
  7. Duration greater than 3 months.
  8. Bibasilar, inspiratory crackles.

Exclusion Criteria:

* under the age of 50
* history of hypersensitivity to interferons
* history of hypersensitivity to biological products such as vaccines
* pregnant or lactating women
* women of child bearing age not pregnancy protected during the study
* unresolved serious cardiovascular disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2000-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Jumper, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical clinic
Groups:
- Interferon Alpha: Treatment with low dose oral interferon alpha lozenges taken 3 times daily (approximately 6 hours apart). Lozenge is to be dissolved under tongue or by moving around in mouth.
Period: Overall Study
Arm/Group | Interferon Alpha
Started | 18
Completed | 11
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Death | 3
Not completed — Non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Interferon Alpha
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 67 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Minimal/no Progression (1 yr) by High Resolution Computed Tomography (HRCT) & Pulmonary Function
Description: Disease progression was determined by comparing results of the High Resolution Computed Tomography(HRCT) and pulmonary function at one year to the baseline HRCT & pulmonary function. The same radiologist did the comparsion for all subjects.
Time Frame: 1 yr
Measure: Number; unit: Participants
Arm/Group | Interferon Alpha
Number analyzed (Participants) | 18
Participants | 12

2. Primary Outcome: Minimal/no Change in Quality of Life
Time Frame: 12 months
Population: Analysis was performed only on those subject who continue on medication for at least one year.
Measure: Number; unit: Participants
Arm/Group | Interferon Alpha
Number analyzed (Participants) | 18
Participants | 12

3. Secondary Outcome: Participants With Change in Cough
Description: changes in cough status after treatment for 1 month.
Time Frame: 1 month
Population: During the course of the study it was noted that subjects experienced a change in the cough that is sometimes associated with IPF. The 6 subjects still enrolled in the study were asked to complete a questionnare regarding the status of the cough.
Measure: Number; unit: Participants
Arm/Group | Interferon Alpha
Number analyzed (Participants) | 6
Participants | 5

ADVERSE EVENTS:
Arm/Group | Interferon Alpha
Serious Adverse Events (participants affected / at risk) | 4/18
Other Adverse Events (participants affected / at risk) | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Alpha (N=18)
Death (Respiratory, thoracic and mediastinal disorders) | 4 (4) — The deaths that occurred were complications of the disease (IPF), not related to the study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No